CLINICAL TRIAL: NCT05866510
Title: A Multicenter, Single-arm, Exploratory Clinical Study of Utidelone Combined With Anlotinib in Advanced Recurrent Metastatic Esophageal Cancer That Has Failed Standard First-line Therapy
Brief Title: Utidelone and Anlotinib in Advanced Recurrent Metastatic Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Beijing Biostar Pharmaceuticals Co., Ltd. (Industry); Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022YJZ92
Record Dates: First submitted 2023-05-07; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Squamous Cell Carcinoma, Utidelone, Anlotinib
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Utidelone and Anlotinib (Experimental): The treatment group will be treated with Utidelone and Anlotinib until the presence of progressive disease or unacceptable toxicity.
  Interventions: Drug: Utidelone and anlotinib

INTERVENTIONS:
Drug: Utidelone and anlotinib — Pretreatment: diphenhydramine 40 mg by intramuscular injection or oral administration, and dexamethasone10 mg and cimetidine 300 mg by intravenous injection 30 minutes prior to Utidelone iv drip at the first day of each cycle.
  Utidelone will be given at 30 mg/m2/d administered intravenously on days 1-5 and Anlotinib 8mg/d took orally on days 1-14 every 21 days.

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerance and efficacy of Utidelone combined with Anlotinib in patients with Advanced or Recurrent Esophageal Carcinoma who failed Standard first line therapy.

DETAILED DESCRIPTION:
Patients with advanced or recurrent esophageal carcinoma who failed standard first-line therapy have a low survival prognosis. There are few treatment options available and the clinical need is great.

The aim of this study is to evaluate the efficacy and safety of Utidelone combined with Anlotinib in patients with Advanced or Recurrent Esophageal Carcinoma who fail first line therapy.

The trial is a single arm design. Patient in the treatment group will accept Utidelone at 30 mg/m2/d administered intravenously on days 1-5 and Anlotinib 8mg/d administered orally on days 1-14, 21 days as one cycle.

Before the use of utidelone, all patients will accept pretreatment: diphenhydramine 40 mg by intramuscular injection or oral administration, and dexamethasone10 mg and cimetidine 300 mg by intravenous injection 30 minutes prior to Utidelone iv drip at the first day of each cycle.

Tumor assessments will be performed at baseline and every 6 weeks (±7 days) after enrollment and will continue until disease progression according to RECIST v1.1 criteria. For patients with no disease progression, tumor evaluation will continue regardless of treatment discontinuation unless the patient begins new antitumor therapy or withdraws informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Histological and/or cytology confirmed advanced or unresectable recurrent esophageal carcinoma
2. All patients had failed first-line chemotherapy (disease progression or unacceptable toxicity occurs).

   Patients may also be included if they receive standard neoadjuvant/adjuvant chemotherapy and relapse within 6 months of completion.
3. All patients were not accepted any treatment(chemotherapy, radiotherapy, surgery, etc.) within 4 weeks before enrollment.
4. The subject has at least one evaluable lesion (measurable or non-measurable) by the RECIST 1.1.
5. Male or female, ≥ 18 years of age, ≤ 75 years of age.
6. ECOG performance status 0-1.
7. Patients with a life expectancy of more than 3 months.
8. Baseline routine blood tests within 1 week prior to enrollment is normal. No rhG-CSF use and no blood transfusion/EPO etc. within 14 days prior to enrollment.

   * Neutrophil count (ANC) ≥ 1.5 × 109/L.
   * Hemoglobin ≥9.0 g/dL.
   * platelet count (PLT) ≥ 80 × 109/L
9. Blood biochemistry test result is normal within 1 week prior to enrollment (based on normal values at each site's laboratory).

   * Total bilirubin (TBIL) ≤ 1.5× the upper limit of normal value (ULN)
   * Serum Glutamic Pyruvic Transaminase/Alanine Amino transferase (SGPT /ALT) ≤ 3× ULN (in the case of liver metastases ≤ 5 × ULN)
   * Serum Glutamic-oxaloacetic Transaminase/Aspartate Aminotransferase (SGOT /AST) ≤ 3× ULN (in the case of liver metastases ≤ 5 × ULN)
   * Creatinine clearance (Ccr) ≥50 ml/min.
10. Fertile males and females of childbearing potential must agree to use effective contraception during the study and within 90 days after the last dose. The blood or urine pregnancy test for female patients of childbearing age prior to enrollment must be negative.
11. Patients must sign the informed consent form and commit to complying with the requirements of this study.

Exclusion Criteria:

1. Patients who have received antitumor therapy, including chemotherapy, radiotherapy, biologic therapy, targeted therapy, immunotherapy, or antitumor herbal therapy, within 4 weeks. With the exception of the following:

   * Nitrosoureas or mitomycin C within 6 weeks prior to the first use of the study drug;
   * Oral fluorouracil and small molecule targeted drugs for 2 weeks prior to the first use of the study drug or within the drug's 5 half-life (whichever is longer);
   * Chinese medicines with antitumor indications within 2 weeks before the first use of the study drug.
2. Major organ surgery (excluding puncture biopsy) within 4 weeks prior to the first dose of study drug had major organ surgery (excluding puncture biopsy) or significant trauma within 4 weeks prior to the first dose of study drug, or required elective surgery during the trial.
3. Patients with symptomatic peripheral neuropathy with CTCAE 5.0 grade ≥2
4. Previous grade 3 or higher neurological related adverse reactions with anti-microtubule drugs.
5. Severe allergy to castor oil, or serious adverse effects from previous use of anti-microtubule drugs Those with severe allergy to castor oil or those who have experienced serious adverse reactions to previous anti-microtubule drugs.
6. Patients who are pregnant (positive result from the pregnancy test) or lactating.
7. Patients whose prior adverse reactions to anti-tumor therapy have not recovered to CTCAE 5.0 grade ≤1 (except for toxicity such as alopecia which poses no safety risk in the judgment of the investigator).
8. Patients with symptomatic CNS metastases or meningeal metastases, or uncontrollable metastases.
9. Patients with an active infection that currently requires systemic anti-infective therapy, including but not limited to: HIV, active hepatitis B/C infection.
10. Patients with history of severe cardiovascular disease
11. Patients with mental disorders or poor compliance.
12. Subjects who, in the opinion of the investigator, have a history of other serious systemic diseases, or other reasons that make participation in this trial inadvisable.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 in all participants | Up to 1 year
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1. For this analysis, ORR will be assessed in all participants who receive at least 1 dose of utidelone and/or anlotinib.

SECONDARY OUTCOMES:
progression-free survival (PFS) per RECIST 1.1 in all participants | Up to 1 year
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 or death due to any cause, whichever occurs first. For this analysis, PFS will be assessed in all participants who receive at least 1 dose of utidelone and/or anlotinib.
duration of response (DOR) per RECIST 1.1 in all participants who achieve partial response (PR) or complete response (CR) | Up to 1 year
  DOR is defined as the interval from response initiation (when either CR or PR is first determined) to progression or death, whichever occurs first.
Overall survival (OS) in all participants | Up to 2 years
  OS is defined as the time from randomization to death due to any cause. For this analysis, OS will be assessed in all participants who receive at least 1 dose of utidelone and/or anlotinib.
Incidence of Treatment-Related Adverse Events | Until 30 days after the last dose of treatment
  An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. The number of participants who experienced ≥1 AE will be presented.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The First Affiliated Hospital of Xinxiang Medical University, Weihui, Henan
  - Suining Central Hospital, Suining, Sichuan
  - Beijing Cancer Hospital, Beijing, China, Beijing

IPD SHARING:
Plan to Share IPD: No